CLINICAL TRIAL: NCT00697489
Title: Pelvic Organ Prolapse Correction Plus Preventive Treatment of Urinary Stress Incontinence vs. Correction of Pelvic Organ Prolapse Followed by Treatment of Urinary Stress Incontinence
Brief Title: Treatment of Urinary Stress Incontinence During or Following Correction of Pelvic Organ Prolapse
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2008
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Urinary incontinence; Mesh
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): unique surgery
  Interventions: Procedure: correction of POP plus preventive continence procedure
- 2 (Active Comparator): Double surgery
  Interventions: Procedure: POP surgery followed by eventual incontinence procedure

INTERVENTIONS:
Procedure: correction of POP plus preventive continence procedure
  Arms: 1
Procedure: POP surgery followed by eventual incontinence procedure
  Arms: 2

SUMMARY:
The incidence of pelvic organ prolapse (POP) in parous women is estimated over 50%. A variety of urinary, bowel and sexual symptoms may be associated with POP. Moreover, a proportion of women who underwent a surgical correction of POP may occur post-surgical urinary incontinence and, thus, if this last presents as genuine stress-type or mixed-type, a second surgical intervention may be required. At this proposal, with the aim to reduce the incidence of postoperative urinary incontinence, the addition of a preventive continence procedure to a POP repair intervention has been widely proposed, but the potential benefits needs to be balanced against potential disadvantages.

Based on these considerations, the aim of this trial will be to compare two different surgical strategies for women with POP without urinary stress incontinence. Specifically, the efficacy to associate and to follow a preventive continence procedure to the correction of POP will be compared.

DETAILED DESCRIPTION:
Women with POP not associated to urinary stress incontinence will be enrolled and randomized in two arms(groups A and B). Patients of group A will be treated with unique surgery (correction of POP plus preventive continence procedure), whereas in patients of group B POP will be surgically corrected and, in case of stress or mixed postoperative incontinence, a further intervention for urinary stress incontinence will be tailored.

All patients eligible will undergo baseline assessment consisting of anthropometric, clinical, hormonal, ultrasonographic and urodynamic evaluations. During the study, the clinical outcomes, and the adverse experience will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic organ prolapse stage 2-3
* Absence of subjective urinary stress incontinence

Exclusion Criteria:

* pregnancy
* <12 months postpartum
* systemic disease known to affect bladder function
* current chemotherapy or radiation therapy
* urethral diverticulum, augmentation cytoplasty, or artificial sphincter
* recent pelvic surgery
* patient age under 18 and over 80
* any previous pelvic surgery, diabetes mellitus and collagen disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
efficacy (cure rate) | 12 months

SECONDARY OUTCOMES:
intra-operative complication rate | one day
postoperative complications rate | 12 months
sexual function | 12 months
quality of life | 12 months
Failure rate | 12 months
Recurrence rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Fulvio Zullo, MD, Study Chair — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Catanzaro, Italy